CLINICAL TRIAL: NCT00049465
Title: Multi-Site Randomized Clinical Trial Comparing Standard Recovery Preparation to Extended Recovery Preparation to Enhance Long Term Function After Marrow or Stem Cell Transplant
Brief Title: Standard Follow-up Compared With Extended Follow-up in Treating Patients Who Have Undergone Stem Cell Transplantation for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: 1430.00; FHCRC-1430.00; NCI-H02-0096; CDR0000258109 (Registry Identifier: PDQ)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Cancer
Keywords: depression; fatigue; menopausal symptoms; transitional care planning; psychosocial effects of cancer and its treatment; accelerated phase chronic myelogenous leukemia; chronic idiopathic myelofibrosis; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; meningeal chronic myelogenous leukemia; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; ovarian choriocarcinoma; ovarian embryonal carcinoma; ovarian yolk sac tumor; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; ovarian polyembryoma; ovarian mixed germ cell tumor; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage II ovarian epithelial cancer; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Burkitt lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III ovarian epithelial cancer; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV ovarian epithelial cancer; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and seminoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma; testicular embryonal carcinoma and seminoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma; testicular teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor; stage III multiple myeloma; chronic eosinophilic leukemia; chronic neutrophilic leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Neoplasms; Depression; Fatigue; Leukemia, Myeloid, Accelerated Phase; Primary Myelofibrosis; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Neuroblastoma; Carcinoma, Ovarian Epithelial; Testicular Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Breast Neoplasms; Carcinoma, Embryonal; Seminoma; Teratoma; Endodermal Sinus Tumor; Teratoma, Testicular; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone | interventions — Therapeutics; Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: fatigue assessment and management
Procedure: management of therapy complications
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Telephone counseling by trained counselors may enhance the well-being and quality of life of patients who have undergone stem cell transplantation for cancer.

PURPOSE: Randomized clinical trial to compare the effectiveness of standard follow-up care with extended follow-up care in treating patients who have undergone stem cell transplantation for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the recovery course of patients with malignancies who undergo standard vs extended recovery preparation after hematopoietic stem cell transplantation.
* Compare the efficacy of these recovery preparations in managing rehabilitation needs, including reduced stamina and cognitive limitations, of these patients.
* Compare the ability of these recovery preparations to assist patients and caregivers in adjusting to unavoidable fluctuations in caregiver roles and emotions.
* Compare the ability of these recovery preparations to assist female patients in managing menopausal symptoms and sexual function changes.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to gender, type of transplantation (allogeneic vs autologous), ethnicity (Caucasian vs non-Caucasian), total body irradiation (yes vs no), and participating center. Patients are randomized to 1 of 2 supportive care arms.

Patients complete 1 baseline assessment prior to transplant and a second assessment after the transplant, approximately 1 week before returning home.

* Arm I (Standard Recovery Preparation): Patients and caregivers receive standard preparation prior to discharge, a booklet of stem cell transplant-related resources and contact information, and the National Cancer Institute-produced publication entitled "Facing Forward".
* Arm II (Recovery Preparation Intervention): Patients and caregivers receive standard preparation and resource materials as in arm I. Women also receive 10 scheduled telephone appointment sessions, lasting 1 hour each, over the first year after returning home. Men receive 9 scheduled telephone appointment sessions in the same manner as the women. The first 5-6 sessions have a specific topic with a corresponding video. The last 4 calls are booster calls to answer questions, identify new problems, and provide support. Patients with acute problems or problems that cannot be handled through regular sessions are referred to the interdisciplinary recovery triage team. Problems addressed by this team include depression, agitation, cognitive change, fatigue, family disruptions, sexuality, and gynecologic or menopausal difficulties.

Patients are followed at 1 and 2 years.

PROJECTED ACCRUAL: A total of 412 patients and their caregivers (385 patients randomized) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a malignancy
* Planned bone marrow, stem cell, or umbilical cord transplantation after a myeloablative conditioning regimen

  * Must have completed radiotherapy and conditioning chemotherapy
  * Must be first stem cell transplantation
  * Must recover sufficiently, physically and cognitively, to be ambulatory and able to live at home
* Must be planning to live with primary caregiver for at least 3 months upon return home
* No refractory breast cancer requiring treatment on a phase I protocol

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Must be able to read, write, and communicate well by phone in English
* Must not be deaf or blind
* Must live in the United States
* Must not be too ill or in too much pain
* No major psychiatric disorders not in remission
* No prisoners
* No prior major alcohol or drug abuse
* No major cognitive problems
* No other concurrent confounding major illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-08; Primary Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Syrjala, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (9):
- United States (9):
  - Stanford University Medical Center, Stanford, California
  - AMC Cancer Research Center, Denver, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington